CLINICAL TRIAL: NCT06113237
Title: Observational Pregnancy Surveillance Program of Patients Exposed to Epidiolex/Epidyolex During Pregnancy to Assess the Risk of Pregnancy and Maternal Complications and Other Events of Interest on the Developing Fetus, Neonate, and Infant
Brief Title: Pregnancy Surveillance Program of Patients Exposed to Epidiolex/Epidyolex During Pregnancy
Status: Recruiting | Type: Observational
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: GWEP21095
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Maternal Complications; Pregnancy Complication; Birth Outcomes, Adverse; Pregnancy
Keywords: Epidiolex; Epidyolex
MeSH Terms: conditions — Pregnancy Complications | interventions — Cannabidiol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Retrospective Pregnancy: Participants who were exposed to at least one dose of Epidiolex/Epidyolex in routine practice during the 13 days prior to last menstrual period (LMP) or at any time during their pregnancy and is no longer pregnant at the time of study enrollment.
  Interventions: Drug: Epidiolex
- Prospective Pregnancy: Participants who were exposed to at least one dose of Epidiolex/Epidyolex in routine practice during the 13 days prior to last menstrual period (LMP) or at any time during their pregnancy and is pregnant at the time of study enrollment.
  Interventions: Drug: Epidiolex

INTERVENTIONS:
Drug: Epidiolex — Oral solution
  Other Names: Epidyolex; Cannabidiol

SUMMARY:
The purpose of this study is to evaluate pregnancy-related health outcomes in participants who are exposed to Epidiolex/Epidyolex during pregnancy and their infant up to 12 months of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with exposure to at least 1 dose of Epidiolex/Epidyolex during the 13 days prior to their LMP or at any time during pregnancy.
2. Verbal or written informed consent to participate

Exclusion criteria:

1) Patients exposed to a non-regulatory approved product containing Cannabidiol (CBD) during pregnancy who do not also have exposure to Epidiolex during the 13 days prior to their LMP or during the pregnancy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who were exposed to at least one dose of Epidiolex/Epidyolex during the 13 days prior to last menstrual period (LMP) or at any time during their pregnancy.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2033-08-31 (Estimated); Study Completion 2033-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of MCM | Up to 12 months post birth
  Rate of Major congenital malformation (MCM) identified in the developing neonate and infant through 12 months of age

SECONDARY OUTCOMES:
Rate of pregnancy outcomes | Up to 10 months gestation
  Rate of the following pregnancy outcomes:
  1. Spontaneous abortion
  2. Elective or therapeutic abortion
  3. Fetal death/stillbirth
  4. Molar or ectopic pregnancy
  5. Preterm delivery
  6. Live birth
Rate of other events of interest in the developing neonate and infant | Up to 12 months post birth
  Rate of the following other events of interest in the developing neonate and infant:
  1. Hospitalizations for serious illness
  2. Medications
  3. Growth and development milestones
  4. Neonatal or infant mortality
  5. Inherited epilepsy syndrome
Rate of maternal complications during pregnancy | Up to 10 months gestation
  Rate of the following maternal complications during pregnancy:
  1. Premature rupture of membranes (PROM)
  2. Pre-eclampsia
  3. Severe pregnancy-induced hypertension
  4. Proteinuria
  5. Gestational diabetes
  6. Intrauterine growth restriction (IUGR)
  7. Measures of fetal growth deficiency (small for gestational age)

CONTACTS AND LOCATIONS:
Locations (1):
- United Biosource LLC, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No